CLINICAL TRIAL: NCT04035278
Title: A Phase 1, Double Blind, Randomized, Placebo-controlled Study to Evaluate the Safety and Immunogenicity of Dengusiil in Healthy Adults
Brief Title: A Phase 1 Safety Study of Dengusiil in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Collaborators: PPD Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dengusiil-01
Record Dates: First submitted 2019-07-25; First posted 2019-07-29 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Prevention of Dengue Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dengusiil (Experimental)
  Interventions: Biological: Dengusiil
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Dengusiil — Dengusiil is provided as lyophilized powder to be reconstituted with 0.5 mL sterile water for injection (sWFI).The reconstituted vaccine is injected as a single 0.5 mL subcutaneous (SC) dose.
  Other Names: Live attenuated tetravalent vaccine containing all four dengue virus serotypes (DENV1, 2, 3 and 4)
  Arms: Dengusiil
Biological: Placebo — Placebo is supplied as a vial of lyophilized powder containing all the components of the vaccine except dengue virus serotypes (DENV1, 2, 3 and 4) to be reconstituted with 0.5 mL sterile water for injection (sWFI).The reconstituted product is injected as a single 0.5 mL subcutaneous (SC) dose.
  Other Names: Lyophilized powder containing all the components of the vaccine except DENV serotypes 1, 2, 3 and 4
  Arms: Placebo

SUMMARY:
This is a Phase 1 study to assess safety and tolerability of a single subcutaneous dose of Dengusiil in healthy adults of 18 to 45 years of age. In this study, immune response to Dengusiil will also be assessed over a period of 6 months and vaccine viremia will also be assessed over a period of 12 days after administration of vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18-45, men, or women.
2. Seronegative for Dengue NS1 and IgM at screening indicating no current dengue infection
3. Seronegative for dengue IgG at screening
4. Participants who are willing to comply with the requirements of the study protocol and attend scheduled visits.
5. Participants who give written informed consent approved by the Human Research Ethics Committee (HREC) governing the site.
6. Participants must have the laboratory parameters within normal range.
7. Participants with Body Mass Index (BMI) between 18 to 30 (both inclusive)
8. Satisfactory baseline medical assessment as assessed by physical examination and normal laboratory values or minor variations those are acceptable for study entry.
9. Participants should agree to not:

   1. donate blood for the purpose of blood transfusion
   2. donate an organ for the purpose of transplantation
   3. to share needles with other people
   4. allow their blood to come in contact with another person's mucous membranes for 84 days post-vaccination.

Exclusion Criteria:

1. Previous dengue vaccination.
2. Presence of acute infection in the preceding 14 days or presence of a temperature ≥ 38.0°C, or acute symptoms of infection greater than of "mild" severity on the scheduled date of first dosing
3. Evidence of any other significant active haematological disease, or having donated > 450 mL of blood within the past three months.
4. Evidence or history of substance abuse including alcohol or previous substance abuse within the last year.
5. Participation or planned participation in a study involving the administration of an investigational compound within the past one month or during this study period.
6. Planned administration of any vaccine not foreseen by the study protocol 4 weeks before and after dosing.
7. History of allergic disease, allergic reactions or known hypersensitivity to any component of the study vaccines.
8. Confirmed or suspected immunosuppressive or immune-deficient condition.
9. A family history of congenital or hereditary immunodeficiency.
10. Chronic administration (defined as more than 14 days) of immune-suppressants or other immune-modifying agents within six months prior to administration of study vaccine. (For corticosteroids, this means prednisone, or equivalent, ≥ 0.5 mg/kg/day; topical or inhalable steroids are allowed.)
11. Laboratory confirmed infection with either hepatitis B virus (HBs Ag positive), hepatitis C virus (anti-HCV positive), or human immunodeficiency virus (HIV) at screening.
12. Known bleeding disorders.
13. Administration of immunoglobulins and/or any blood products within the three months preceding the administration of study vaccines or planned administration during the study period.
14. Women who are pregnant, breast-feeding, or considering becoming pregnant.
15. Any other condition, which in the opinion of the investigator, might interfere with the study objectives, jeopardize the safety or rights of the participant or making it unlikely the participant could complete the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Solicited local and systemic reactions | 21 days
Occurrence, severity, and relatedness to vaccination of unsolicited adverse events | 21 days
Occurrence, severity, and relatedness to vaccination of serious adverse events | 180 days
Proportion of participants with clinically significant abnormal safety laboratory (hematology and chemistry parameters) findings | 8 days
Proportion of participants with clinically significant physical examination and vital signs findings | 180 days

SECONDARY OUTCOMES:
Proportion of participants with seroconversion for DENV-1 to 4 virus neutralization antibodies (PRNT50) titer | 84 days
The percentage of participants seropositive for DENV-1 to 4 virus neutralizing antibodies | 84 days
The percentage of participants seropositive for DENV-1 to 4 virus neutralizing antibodies | 180 days
Geometric mean titers (GMTs) of DENV-1 to 4 virus neutralization antibodies | 56 days
GMTs of DENV-1 to 4 virus neutralization antibodies | 84 days
Proportion of participants with viremia for each of DENV-1 to 4 | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: PRASAD KULKARNI, MD, Study Director — SERUM INSTITUTE OF INDIA
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gunale B, Farinola N, Yeolekar L, Shrivastava S, Girgis H, Poonawalla CS, Dhere RM, Arankalle V, Chandra Mishra A, Mehla R, Kulkarni PS. A Phase 1, double-blind, randomized, placebo-controlled study to evaluate the safety and immunogenicity of a tetravalent live attenuated dengue vaccine in adults. Vaccine. 2023 Aug 31;41(38):5614-5621. doi: 10.1016/j.vaccine.2023.07.045. Epub 2023 Jul 31. PMID 37532611